CLINICAL TRIAL: NCT02189525
Title: AWARE: Mild Traumatic Brain Injury in Collegiate Athletes - A Prospective Study With Blood-based Biomarkers, Advanced Neuroimaging and the Head Impact Telemetry System (HITS)
Brief Title: Evaluation of Mild TBI in Collegiate Athletes
Acronym: AWARE
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HHC-001
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; sports head injury; sports concussion
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sports induced concussion: Exposure to sports induced concussion
- Routine Athletic Exertion: Exposure to routine athletic exertion without sports-induced concussion (non-concussion control)

SUMMARY:
The purpose of this study is to evaluate blood-based biomarkers before and after sports-induced concussion using neuroimaging and head impact sensor technology.

ELIGIBILITY:
Inclusion Criteria:

1. University of Florida student athlete involved in Men's Football, Men and Women's Basketball, Men and Women's Swimming, Men and Women's Diving, Women's Soccer, or Women's Lacrosse or University of Florida student athlete not participating in those sports who is being treated for a sports-related head injury.
2. Age greater than or equal to 18 years of age.
3. Willing to undergo the Informed Consent Process and provide Informed Consent prior to enrollment into the study.

Exclusion Criteria:

* Subject is otherwise determined by the Investigator to be medically unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Collegiate atheltes from University of Florida involved in Men's Football, Women's Soccer, or Women's Lacrosse
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-08; Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Correlation of serum biomarker levels with neuroanatomic and neuropathologic changes from baseline using neuroimaging, following sports-related concussion | Baseline and up to 48 months

SECONDARY OUTCOMES:
Correlation of serum biomarker levels with head acceleration data using head impact telemetry system following sports-related concussion | Baseline and up to 48 months
Correlation of serum biomarker levels and neuroimaging results to standard clinical measures of concussion in the acute phase of injury and at the completion of collegiate athletic participation | Baseline and up to 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Asken BM, Bauer RM, DeKosky ST, Houck ZM, Moreno CC, Jaffee MS, Weber AG, Clugston JR. Concussion Biomarkers Assessed in Collegiate Student-Athletes (BASICS) I: Normative study. Neurology. 2018 Dec 4;91(23):e2109-e2122. doi: 10.1212/WNL.0000000000006613. Epub 2018 Nov 7. PMID 30404785
- [Background] Asken BM, Bauer RM, DeKosky ST, Houck ZM, Moreno CC, Jaffee MS, Dubose DN, Boone JK, Weber AG, Clugston JR. Concussion BASICS II: Baseline serum biomarkers, head impact exposure, and clinical measures. Neurology. 2018 Dec 4;91(23):e2123-e2132. doi: 10.1212/WNL.0000000000006616. Epub 2018 Nov 7. PMID 30404782
- [Background] Asken BM, Bauer RM, DeKosky ST, Svingos AM, Hromas G, Boone JK, DuBose DN, Hayes RL, Clugston JR. Concussion BASICS III: Serum biomarker changes following sport-related concussion. Neurology. 2018 Dec 4;91(23):e2133-e2143. doi: 10.1212/WNL.0000000000006617. Epub 2018 Nov 7. PMID 30404786